CLINICAL TRIAL: NCT06140875
Title: Amplitude Modulated Radiofrequency Electromagnetic Field Treatment Combined With Radiochemotherapy and Maintenance Chemotherapy in Patients With Glioblastoma (Brain-RF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Pirus Ghadjar, Prof. Dr., Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Brain-RF
Record Dates: First submitted 2023-11-15; First posted 2023-11-20 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Radiochemotherapy (RCT) and maintenance chemotherapy (CT) according to Stupp et al. 2005 combined with radiofrequency electromagnetic field treatment.
  The standard therapy involves gross- or subtotal tumor resection if feasible (alternatively biopsy only) followed by RCT (60 Gy over six weeks) with concomitant CT (temozolomide 75mg/m2) on all days, followed by maintenance CT (temozolomide150-200 mg/m2) on d1-5 for six cycles every 28 days.
  The trial intervention includes radiofrequency electromagnetic field treatment for 60 minutes three times a week during RCT and twice a week during d1-5 of maintenance CT, resulting in a total number of 30 radiofrequency electromagnetic field treatment therapy sessions.
  Interventions: Device: Radiofrequency electromagnetic field treatment

INTERVENTIONS:
Device: Radiofrequency electromagnetic field treatment — Radiofrequency electromagnetic field treatment using a carrier frequency of 13.56 MHz
  Other Names: mEHT; capacitive hyperthermia; electrohyperthermia

SUMMARY:
Combined chemoradiation and radiofrequency electromagnetic field treatment for patients with glioblastoma

DETAILED DESCRIPTION:
Charité Universitätsmedizin Berlin is currently the only German University Hospital with an available capacitive radiofrequency electromagnetic field treatment device. While there is retrospective data available regarding the assumed effectiveness and low toxicity profile of radiofrequency electromagnetic field treatment for glioblastoma in the palliative setting, there is only few prospective data available on the combined effect first-line chemoradiation and radiofrequency electromagnetic field treatment. The investigators aim to conduct a feasibility trial and plan to compare the results with data of a prospective trial with a comparable patient population.

ELIGIBILITY:
Inclusion Criteria:

* Pathological evidence of newly diagnosed glioblastoma according to WHO classification criteria
* Patients 18 to 70 years of age with a WHO performance status of 2 or less
* All patients must sign written informed consent
* Adequate hematologic, renal, and hepatic function (absolute neutrophil count, ≥1,5 x 103/μL; platelet count, ≥100 x 103/μL; serum creatinine ≤1.7 mg/dL; total bilirubin > upper limit of normal; AST or ALT ≤3 times the upper limit of normal)
* Patient must have received subtotal or gross total resection of the tumor
* MGMT-promotor methylated patients must have refused therapy according to the CeTeG/NOA-09 protocol (+ Lomustin)
* Patient must be planned for concomitant RCT with a total RT dose of 60 Gy over six weeks and temozolomide followed by six cycles of maintenance CT using temozolomide

Exclusion Criteria:

* Previous cranial RT
* Cytostatic therapy / anti-angiogenic substances / CT or radiation therapy for cancer within the past 5 years
* History of cancers or other comorbidities that limit life expectancy to less than five years
* Postoperative evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness)
* Technical impossibility to use magnetic resonance imaging (MRI) or known allergies against MRI and/or computed tomography (CT) contrast agents
* Technical impossibility to use AM-RF-EMF (pacemaker, defibrillator or deep brain stimulator, metal implants)
* Participants of childbearing age unwilling to use or not capable of using effective contraception
* Pregnant patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2029-05-14 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
PFS at 6 months | 6 months after surgery or biopsy
  Progression-free survival

SECONDARY OUTCOMES:
OS | Through study completion, an average of 15 months
  Overall Survival
Acute and late toxicity | During 5,5 years of trial conduction
  CTCAE version 5
Subsequent salvage treatment of the brain | During 5,5 years of trial conduction
  Need for brain surgery, new drug therapy or additional radiotherapy of the brain
PFS | During 5,5 years of trial conduction
  Progression-free survival
QOL | During 5,5 years of trial conduction
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-BN20
Mini mental state examination | During 5,5 years of trial conduction
  Brain function testing
QOL | During 5,5 years of trial conduction
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30
Depression and anxiety testing | During 5,5 years of trial conduction
  Hospital Anxiety and Depression Scale (HADS-D)

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided